CLINICAL TRIAL: NCT05572216
Title: A CCafU-UroCCR Randomized Trial: 3D Image-Guided Robot-AssisTEd Partial Nephrectomy for Renal Complex Tumor (UroCCR N°99)
Acronym: ACCURATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EssaiClinique_ACCURATE
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Renal Tumor; Renal Cancer
Keywords: image guidance; augmented reality; robotics
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Intervention Model Description: ACCURATE is a nation-wide, single-blind, multicentric, prospective randomized controlled trial enrolling patients with a single complex renal mass, defined as RENAL NS≥7. Randomization (1:1) between the experimental and the conventional group will take place on day of inclusion and will be stratified by center.
Who Masked: Participant
Masking Description: single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional group (No Intervention): Robot-Assisted Partial Nephrectomy without 3D navigation
- 3D IGRAPN GROUP (Experimental): Robot-Assisted Partial Nephrectomy with 3D navigation
  Interventions: Procedure: Robot assisted partial nephrectomy with 3D image guidance

INTERVENTIONS:
Procedure: Robot assisted partial nephrectomy with 3D image guidance — patient have a partial nephrectomy for renal complex tumor
  Other Names: without 3D image guidance
  Arms: 3D IGRAPN GROUP

SUMMARY:
The goal of this clinical trial is to evaluate peri and post-operative outcomes as well as long-term survival of 3D IGRAPN compared to conventional Robot-Assisted Partial Nephrectomy (RAPN) for moderate and highly complex renal tumors.

The main questions aim to answer:

* peri-operative complications
* oncological safety
* long term renal function Participants will be asked to do undergo 3D-IGRAPN. Researchers will compare 3D-IGRAPN to RAPN to see if peri-operative outcomes are better in the experimental group.

DETAILED DESCRIPTION:
Robot-assisted partial nephrectomy (RAPN) is the standard treatment for localized kidney tumors. New 3D modeling and reconstruction technologies have enabled the development of real time imageguided surgery using virtual reality (VR). In view of advances in artificial intelligence and surface recognition based on deep-learning, augmented reality (AR) by merging a 3D reconstructed virtual image onto the real per-operative view represents the next step in image-guided surgery.

3D IG-RAPN using Synapse 3D (Fujifilm) and DaVinci Tile-Pro display (Intuitive Surgical) vs conventional RAPN without 3D navigation in 12 high-volume urological centers from the UroCCR Network.

Outcoume : Primary endpoint is a composite validated score (TRIFECTA) evaluating peri-operative complications as well as oncological safety and long-term renal function preservation. Secondary endpoints assess long-term survival, ergonomics and surgeon satisfaction. A medico-economic evaluation will be performed.

Methodology: ACCURATE is a nation-wide, single-blind, multicentric, prospective randomized controlled trial enrolling 694 patients with a single complex renal mass, defined as RENAL NS≥7.

Randomization (1:1) between the experimental and the conventional group will take place on day of inclusion and will be stratified by center.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Indication of RAPN for suspicious renal tumor
* Moderate or high complexity renal tumor (RENAL Nephrometry Score (NS) >7)
* Da Vinci® surgical system available for the surgery
* Patient affiliated to the French social security system or an equivalent system
* Signed informed consent form UroCCR and ACCURATE

Exclusion Criteria:

* Medical contraindication to RAPN
* Renal insufficiency forbidding iodine injection
* Patient with allergy to iodinated contrast products
* Patient concerned by articles L1121-5 to 8 of the French public health code (protected persons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 694 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
TRIFECTA score | 1 month
  evaluating peri-operative outcome complications as well as oncological safety and long-term renal function preservation.

SECONDARY OUTCOMES:
Recurrence free survival | 2 and 5 years
  Recurrence-free survival and Overall survival
Overall survival | 2 and 5 years
  Overall Survival
Number of Conversion to radical nephrectomy | Intraopertively
  Need to convert to radical nephrectomy for intra-operative reasons
rate of Off clamp or superselective ischemia | Intraoperatively
  use of techniques without renal artery clamping
Amount of parenchyma preserved (according to CT scan) | Month 6
  Preservation of safe kidney
Blood loss | Intra-operatively
  Blood loss
NASA TLX | at the end of the surgery
  Ergonomy score (questionnaire completed at the end of the procedure by the surgeon)
Warm ischemia time | Intra-operatively
  Warm ischemia time
Medico-economic evaluation | Month 1 and 6
  ncremental cost-utility ratio (ICUR) expressed as the extra cost per a QALY gained by the 3D-IGRAPN strategy compared to standard RAPN.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc DESCOTES, Pr, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - University Hospital Grenoble, Grenoble
  - university HospitalGrenoble, Grenoble

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michiels C, Khene ZE, Prudhomme T, Boulenger de Hauteclocque A, Cornelis FH, Percot M, Simeon H, Dupitout L, Bensadoun H, Capon G, Alezra E, Estrade V, Bladou F, Robert G, Ferriere JM, Grenier N, Doumerc N, Bensalah K, Bernhard JC. 3D-Image guided robotic-assisted partial nephrectomy: a multi-institutional propensity score-matched analysis (UroCCR study 51). World J Urol. 2023 Feb;41(2):303-313. doi: 10.1007/s00345-021-03645-1. Epub 2021 Apr 2. PMID 33811291
- [Background] Porpiglia F, Checcucci E, Amparore D, Piramide F, Volpi G, Granato S, Verri P, Manfredi M, Bellin A, Piazzolla P, Autorino R, Morra I, Fiori C, Mottrie A. Three-dimensional Augmented Reality Robot-assisted Partial Nephrectomy in Case of Complex Tumours (PADUA >/=10): A New Intraoperative Tool Overcoming the Ultrasound Guidance. Eur Urol. 2020 Aug;78(2):229-238. doi: 10.1016/j.eururo.2019.11.024. Epub 2019 Dec 30. PMID 31898992
- [Background] Long JA, Fiard G, Giai J, Teyssier Y, Fontanell A, Overs C, Poncet D, Descotes JL, Rambeaud JJ, Moreau-Gaudry A, Ittobane T, Bouzit A, Bosson JL, Lanchon C. Superselective Ischemia in Robotic Partial Nephrectomy Does Not Provide Better Long-term Renal Function than Renal Artery Clamping in a Randomized Controlled Trial (EMERALD): Should We Take the Risk? Eur Urol Focus. 2022 May;8(3):769-776. doi: 10.1016/j.euf.2021.04.009. Epub 2021 Apr 27. PMID 33931361